CLINICAL TRIAL: NCT01322672
Title: Peri-Anesthetic Imaging Compared With Neurocognitive Testing: A Pilot Study
Brief Title: Peri-Anesthetic Imaging of Cognitive Dysfunction
Acronym: PAICOD
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James L. Blair, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: IRB#100885
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Cognitive Dysfunction; Delirium; Dementia; Neurotoxicity
Keywords: Anesthetic Agents; POCD; Delirium; Cognitive Testing; Aging; Surgery; fMRI; Diffusion Tensor Imaging; White Matter
MeSH Terms: conditions — Postoperative Cognitive Complications; Delirium; Dementia; Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent data suggests that anesthetics can have prolonged effects on gene expression, protein synthesis and processing as well as cellular function in ways that the investigators are only beginning to understand, especially in the very young and the elderly. Within moments to days of emerging from anesthesia - cardiac or non-cardiac - some patients experience mild to very severe disorientation and changes in memory and thinking ability without apparent cause. For the vast majority of patients, this Post-Operative Cognitive Dysfunction (POCD), generally subsides, but for some with "diminished cognitive reserve" - especially the elderly, those with less education or prior CNS events such as stroke or early dementia - changes in memory and executive function may persist. If prolonged for more than three months, POCD has been linked to an increased risk of death. In 1-2% of elderly patients, the problem may ultimately continue for more than a year, leading to a loss of ability to care for themselves and early demise. Though this may seem like a small percentage, seniors will comprise up to 40% of the 50-75 million surgical procedures performed annually over the next 20-30 years. This amounts to 70,000 - 200,000 elder affected, and for them and their families, the cost of POCD in longer-term care, lost wages, and extended suffering will remain very high.

DETAILED DESCRIPTION:
For more than 160 years, "modern" anesthesia has provided immense benefit to patients of all ages. However, over the past several years, concern has been growing that for patients at the extremes of age, some anesthetic agents may harbor subtle, previously minimally examined, serious neurotoxic effects which can cause lasting decline in the function of the central nervous system (CNS). For the elderly, these effects may manifest in lasting post-operative deterioration of memory and the capacity for normal information processing that can result in the inability to perform the activities of daily living (ADLs) with eventual early demise. Unfortunately, even though our ability to evaluate anesthetic risk has grown asymptotically for virtually every organ system, the brain remains neglected. And even though we know a good deal about effect sites for general anesthetic agents, we still have an incomplete understanding of the potential toxic effects of anesthetics on the brain. Therefore, employing a human surgical model (endoscopic prostatectomy), we propose a pilot study of 15 otherwise neurologically intact, ASA I - III, males, 65+ year of age. After pre-enrollment screening (MMSE & BDI) and standard pre-op evaluation, subjects will undergo both anatomic and functional MRI studies plus a battery of neurocognitive tests (NCT) at two time points approximately 2-3 weeks apart prior to surgery. These pre-op studies will establish both a "non-surgical control" for the study as well as a baseline for post-op studies. 2-3 weeks after surgery, MRI and NCT will be repeated. The study aims to determine if MRI can demonstrate changes in the CNS pre-op vs post-op that relate to anesthesia and surgery and how those changes might correlate with NCT over the same interval.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+ years; ASA I - III; capable and willing to consent
* Scheduled for 3+ hour Endoscopic Prostatectomy under general anesthesia
* Baseline MMSE > 20 (exclude dementia)
* All suitable for MRI testing

Exclusion Criteria:

* Hx Autoimmune Disease
* Severe visual or auditory disorder/handicaps
* Unable to read or understand English
* Pre-existing cognitive impairment; e.g., MS, AD or Parkinson's Disease, etc.
* Patients not expected to be able to complete the 2-3 week postoperative testing
* Major psychiatric condition such as bipolar disorder, schizophrenia
* Severe Panic Disorder
* Any implanted ferrous metal

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects will be non-rheumatoid, non-immune-compromised, males and females, 65+ years old, scheduled for open abdominal surgery under general anesthesia of 3+ hour's duration.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Comparison of preoperative vs postoperative Brain MRI changes | 2 months
  Anesthetics can have prolonged effects on gene expression, protein synthesis and processing as well as cellular function, especially in the very young and the elderly. After anesthesia, some patients experience mild to very severe disorientation and even delirium without apparent cause. In the elderly, this Post-Operative Cognitive Dysfunction (POCD) - including changes in memory and executive function may persist and has been linked to an increased risk of death. Over the next 20-30 years, 40% of 65+ year-olds will undergo surgery; the cost of POCD in longer-term care, lost wages, and extended suffering of patients and families will remain high.

SECONDARY OUTCOMES:
Preoperative vs Postoperative Neurocognitive Testing | 2 Months
  Pre- vs postoperative Neurocognitive Testing (NCT) is currently the primary method used to quantify changes in cognitive indices, including memory, processing speed, motor function, etc. This study will compare such pre- and post-op NCT with pre-and post-op MRI and fMRI to determine relationships between changes in each of these modalities.

CONTACTS AND LOCATIONS:
Overall Officials: James L Blair, DO, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Perouansky M, Hemmings HC Jr. Neurotoxicity of general anesthetics: cause for concern? Anesthesiology. 2009 Dec;111(6):1365-71. doi: 10.1097/ALN.0b013e3181bf1d61. No abstract available. PMID 19934883
- [Background] Fudickar A, Peters S, Stapelfeldt C, Serocki G, Leiendecker J, Meybohm P, Steinfath M, Bein B. Postoperative cognitive deficit after cardiopulmonary bypass with preserved cerebral oxygenation: a prospective observational pilot study. BMC Anesthesiol. 2011 Mar 14;11:7. doi: 10.1186/1471-2253-11-7. PMID 21401948
- [Background] Newman S, Stygall J, Hirani S, Shaefi S, Maze M. Postoperative cognitive dysfunction after noncardiac surgery: a systematic review. Anesthesiology. 2007 Mar;106(3):572-90. doi: 10.1097/00000542-200703000-00023. PMID 17325517
- [Background] Shioiri A, Kurumaji A, Takeuchi T, Matsuda H, Arai H, Nishikawa T. White matter abnormalities as a risk factor for postoperative delirium revealed by diffusion tensor imaging. Am J Geriatr Psychiatry. 2010 Aug;18(8):743-53. doi: 10.1097/JGP.0b013e3181d145c5. PMID 20220599
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] Teeling JL, Perry VH. Systemic infection and inflammation in acute CNS injury and chronic neurodegeneration: underlying mechanisms. Neuroscience. 2009 Feb 6;158(3):1062-73. doi: 10.1016/j.neuroscience.2008.07.031. Epub 2008 Jul 25. PMID 18706982
- [Background] Hudetz JA, Patterson KM, Byrne AJ, Pagel PS, Warltier DC. Postoperative delirium is associated with postoperative cognitive dysfunction at one week after cardiac surgery with cardiopulmonary bypass. Psychol Rep. 2009 Dec;105(3 Pt 1):921-32. doi: 10.2466/PR0.105.3.921-932. PMID 20099555
- [Background] Tucker AM, Stern Y. Cognitive reserve in aging. Curr Alzheimer Res. 2011 Jun;8(4):354-60. doi: 10.2174/156720511795745320. PMID 21222591
- [Background] Buckner RL, Andrews-Hanna JR, Schacter DL. The brain's default network: anatomy, function, and relevance to disease. Ann N Y Acad Sci. 2008 Mar;1124:1-38. doi: 10.1196/annals.1440.011. PMID 18400922
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878